CLINICAL TRIAL: NCT06665490
Title: Pilot Study to Characterize the Microbiome in Cutaneous T Cell Lymphoma Skin Lesions Before and After Use of CLn® Skin Care Body Wash
Status: Not yet recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Xiaolong (Alan) Zhou, Principal Investigator, Northwestern University
Other Study IDs: STU00222221
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Cutaneous T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin microbiome swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Mycosis Fungoides patients: Patients with mycosis fungoides will be enrolled at Northwestern Memorial Hospital Dermatology
  Interventions: Other: CLn Body Wash

INTERVENTIONS:
Other: CLn Body Wash — All enrolled patients will self-administer at home the commercially available study product (CLn Body Wash) containing 0.006% NaOCl body wash in a sealed, child-safe pump dispenser to use daily for 8 weeks by wetting the body thoroughly with showering, lathering the study product on the body with special attention to affected areas, leaving on the skin for 2 minutes, and rinsing off with warm water.

SUMMARY:
In this pilot study of patients with mycosis fungoides, the most common form of CTCL, we propose to primarily evaluate the impact of daily use of the CLn Body Wash (dilute sodium hypochlorite (0.006% NaOCl)) on the microbiota of CTCL lesions. Should dilute sodium hypochlorite body wash improve the microbiome of MF, reducing the abundance of S. aureus, future, larger studies can more fully evaluate the impact on pruritus, erythema, scaling, disease evolution and its role in CTCL management.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-89 years of age with active mycosis fungoides.
* Patients with concurrent and prior malignancies are allowed as long as any concurrent malignancy does not directly involve the same skin site.

Exclusion Criteria:

* Patients currently or recently (within past 4 weeks) on topical or systemic antibiotics, pregnant persons, or persons with potential of becoming pregnant or are/will be breastfeeding
* Patients that have initiated a new skin-directed therapy over the past month.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mycosis fungoides (MF) will be enrolled at Northwestern Memorial Hospital Dermatology outpatient clinic at 676 N St. Clair Street, Suite 1600, Chicago, IL 60611.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Reduction of S. aureus skin microbiome | 8 weeks
  Reduction of S. aureus relative abundance between baseline (Week 0) and Week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Zhou, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States